CLINICAL TRIAL: NCT02096861
Title: A Randomized, Double-Blind, Parallel-Group, Phase 3 Study to Demonstrate Noninferiority in Efficacy and to Assess Safety of CT-P13 Compared to Remicade in Patients With Active Crohn's Disease
Brief Title: Demonstrate Noninferiority in Efficacy and to Assess Safety of CT-P13 in Patients With Active Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celltrion (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT-P13 3.4; 2013-004497-10 (EudraCT Number)
Record Dates: First submitted 2014-03-24; First posted 2014-03-26 (Estimated); Results first posted 2018-04-11 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2018-03

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — CT-P13; Infliximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CT-P13 - CT-P13 (Experimental): CT-P13 followed by CT-P13 from Week 30
  Interventions: Biological: CT-P13
- CT-P13 - Remicade (Active Comparator): CT-P13 followed by Remicade from Week 30
  Interventions: Biological: CT-P13; Biological: Remicade
- Remicade - Remicade (Active Comparator): Remicade followed by Remicade from Week 30
  Interventions: Biological: Remicade
- Remicade - CT-P13 (Experimental): Remicade followed by CT-P13 from Week 30
  Interventions: Biological: CT-P13; Biological: Remicade

INTERVENTIONS:
Biological: CT-P13 — CT-P13 (5 mg/kg) by intravenous (IV) infusion administered as a 2 hour IV infusion per dose
  Arms: CT-P13 - CT-P13; CT-P13 - Remicade; Remicade - CT-P13
Biological: Remicade — Remicade (5 mg/kg) by intravenous (IV) infusion administered as a 2 hour IV infusion per dose
  Arms: CT-P13 - Remicade; Remicade - CT-P13; Remicade - Remicade

SUMMARY:
This study is to assess noninferiority in efficacy and to assess overall safety of CT P13 compared to Remicade in patients with active Crohn's disease up to Week 54.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with active Crohn's disease and a Crohn's disease activity index score between 220 and 450 points

Exclusion Criteria:

* Patient who has previously received a biological agent for the treatment of Crohn's disease and/or a Tumor necrosis factor (TNF)-alpha inhibitor for the treatment of other disease.
* Patient who has allergies to any of the excipients of infliximab, any other murine and/or human proteins, or patient with a hypersensitivity to immunoglobulin product.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2014-09-19 (Actual); Primary Completion 2016-01-11 (Actual); Study Completion 2017-02-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nashville Medical Research Institute, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Narula N, Wong ECL, Dulai PS, Marshall JK, Jairath V, Reinisch W. Comparative Effectiveness of Biologics for Endoscopic Healing of the Ileum and Colon in Crohn's Disease. Am J Gastroenterol. 2022 Jul 1;117(7):1106-1117. doi: 10.14309/ajg.0000000000001795. Epub 2022 Apr 15. PMID 35435862
- [Derived] Dulai PS, Wong ECL, Reinisch W, Narula N. Clinical Decision Support Tool for Infliximab in Crohn's Disease. Clin Gastroenterol Hepatol. 2022 May;20(5):e1192-e1195. doi: 10.1016/j.cgh.2021.06.037. Epub 2021 Jun 30. PMID 34216825
- [Derived] Wong ECL, Buffone E, Lee SJ, Dulai PS, Marshall JK, Reinisch W, Narula N. End of Induction Patient-reported Outcomes Predict Clinical Remission but Not Endoscopic Remission in Crohn's Disease. J Crohns Colitis. 2021 Jul 5;15(7):1114-1119. doi: 10.1093/ecco-jcc/jjaa242. PMID 33245751
- [Derived] Ye BD, Pesegova M, Alexeeva O, Osipenko M, Lahat A, Dorofeyev A, Fishman S, Levchenko O, Cheon JH, Scribano ML, Mateescu RB, Lee KM, Eun CS, Lee SJ, Lee SY, Kim H, Schreiber S, Fowler H, Cheung R, Kim YH. Efficacy and safety of biosimilar CT-P13 compared with originator infliximab in patients with active Crohn's disease: an international, randomised, double-blind, phase 3 non-inferiority study. Lancet. 2019 Apr 27;393(10182):1699-1707. doi: 10.1016/S0140-6736(18)32196-2. Epub 2019 Mar 28. PMID 30929895
- [Derived] Husereau D, Feagan B, Selya-Hammer C. Policy Options for Infliximab Biosimilars in Inflammatory Bowel Disease Given Emerging Evidence for Switching. Appl Health Econ Health Policy. 2018 Jun;16(3):279-288. doi: 10.1007/s40258-018-0371-0. PMID 29411318

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CT-P13 - CT-P13 | CT-P13 - Remicade | Remicade - Remicade | Remicade - CT-P13
Started | 56 (CT-P13 followed by CT-P13 from Week 30) | 55 (CT-P13 followed by Remicade from Week 30) | 54 (Remicade followed by Remicade from Week 30) | 55 (Remicade followed by CT-P13 from Week 30)
Drug Switching at Week 30 | 48 | 44 | 41 | 47
Completed | 44 | 40 | 37 | 45
Not Completed | 12 | 15 | 17 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CT-P13 - CT-P13 | CT-P13 - Remicade | Remicade - Remicade | Remicade - CT-P13 | Total
Number analyzed (Participants) | 56 | 55 | 54 | 55 | 220
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1 | 0 | 2
  Between 18 and 65 years | 54 | 53 | 52 | 55 | 214
  >=65 years | 2 | 1 | 1 | 0 | 4
Age, Continuous [Median (Full Range); unit: years] | 39 [19 to 68] | 31 [18 to 69] | 31 [18 to 69] | 35 [19 to 63] | 33 [18 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 21 | 28 | 21 | 97
  Male | 29 | 34 | 26 | 34 | 123
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 11 | 14 | 13 | 16 | 54
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 45 | 41 | 40 | 39 | 165
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 0 | 0 | 0 | 2 | 2
  Brazil | 0 | 1 | 1 | 0 | 2
  Denmark | 1 | 0 | 0 | 0 | 1
  France | 2 | 1 | 1 | 1 | 5
  Germany | 0 | 0 | 1 | 1 | 2
  Hungary | 1 | 5 | 4 | 1 | 11
  Israel | 8 | 6 | 8 | 4 | 26
  Italy | 3 | 4 | 2 | 3 | 12
  Mexico | 2 | 0 | 0 | 2 | 4
  Netherlands | 2 | 0 | 1 | 0 | 3
  Poland | 1 | 1 | 3 | 0 | 5
  Romania | 2 | 1 | 2 | 3 | 8
  Russia | 15 | 15 | 8 | 12 | 50
  South Korea | 11 | 14 | 13 | 16 | 54
  Ukraine | 7 | 6 | 10 | 9 | 32
  United States | 1 | 1 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: The Number and Percentage of Patients Achieving Clinical Response According to Crohn's Disease Activity Index (CDAI)-70 Criteria at Week 6
Description: A patient was defined as having a CDAI-70 response if there was a decrease in CDAI score of 70 points or more at Week 6 comparing to the baseline value.
Time Frame: at Week 6
Population: CT-P13 treatment group including CT-P13 - CT-P13 and CT-P13 - Remicade treatment groups.
  Remicade treatment group including Remicade - Remicade and Remicade - CT-P13 treatment groups.
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P13 | Remicade
Number analyzed (Participants) | 111 | 109
Participants | 77 | 81

2. Secondary Outcome: The Number and Percentage of Patients Achieving Clinical Response According to CDAI-70 Criteria at Week 30
Description: A patient was defined as having a CDAI-70 response if there was a decrease in CDAI score of 70 points or more from the baseline value.
Time Frame: Week 30
Population: CT-P13 group including CT-P13-CT-P13 and CT-P13-Remicade treatment group Remicade group including Remicade-Remicade and Remicade-CT-P13 treatment group
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P13 | Remicade
Number analyzed (Participants) | 111 | 109
Participants | 85 | 82

3. Secondary Outcome: The Number and Percentage of Patients Achieving Clinical Response According to CDAI-70 Criteria at Week 54
Description: as for outcome 2
Time Frame: Week 54
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P13 - CT-P13 | CT-P13 - Remicade | Remicade - Remicade | Remicade - CT-P13
Number analyzed (Participants) | 56 | 55 | 54 | 55
Participants | 44 | 39 | 38 | 42

4. Secondary Outcome: The Number and Percentage of Patients Achieving Clinical Remission at Week 6
Description: Clinical remission was defined as an absolute CDAI score of less than 150 points.
Time Frame: Week 6
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P13 | Remicade
Number analyzed (Participants) | 111 | 109
Participants | 47 | 49

5. Secondary Outcome: The Number and Percentage of Patients Achieving Clinical Remission at Week 30
Description: Clinical remission was defined as an absolute CDAI score of less than 150 points.
Time Frame: Week 30
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P13 | Remicade
Number analyzed (Participants) | 111 | 109
Participants | 61 | 62

6. Secondary Outcome: The Number and Percentage of Patients Achieving Clinical Remission at Week 54
Description: Clinical remission was defined as an absolute CDAI score of less than 150 points.
Time Frame: Week 54
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P13 - CT-P13 | CT-P13 - Remicade | Remicade - Remicade | Remicade - CT-P13
Number analyzed (Participants) | 56 | 55 | 54 | 55
Participants | 35 | 32 | 29 | 33

7. Secondary Outcome: The Short Inflammatory Bowel Disease Questionnaire (SIBDQ)
Description: SIBDQ is scored with 10 sub-question which can be scored from 1 to 7. Therefore, SIBDQ can be scored from 7 to 70.
  Higher values of SIBDQ represent a better patient disease outcome.
Time Frame: Up to Week 30
Population: Number Analyzed at each visit is the number of patients who had SIBDQ score at each visit.
  CT-P13 group including CT-P13-CT-P13 and CT-P13-Remicade treatment group Remicade group including Remicade-Remicade and Remicade-CT-P13 treatment group
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | CT-P13 | Remicade
Number analyzed (Participants) | 111 | 109
scores on a scale
  Baseline | 34.3 (10.92) | 33.9 (9.27)
  Week 6: number analyzed (Participants) | 107 | 107
  Week 6 | 46.4 (10.86) | 45.8 (12.54)
  Week 30: number analyzed (Participants) | 92 | 88
  Week 30 | 51.1 (11.96) | 52.5 (10.68)

8. Secondary Outcome: The Short Inflammatory Bowel Disease Questionnaire
Description: as for outcome 7
Time Frame: Baseline and Week 54
Population: Number Analyzed at each visit is the number of patients who had SIBDQ score at each visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | CT-P13 - CT-P13 | CT-P13 - Remicade | Remicade - Remicade | Remicade - CT-P13
Number analyzed (Participants) | 56 | 55 | 54 | 55
scores on a scale
  Baseline | 34.7 (10.61) | 33.8 (11.31) | 33.3 (9.77) | 34.5 (8.81)
  Week 54: number analyzed (Participants) | 45 | 41 | 37 | 47
  Week 54 | 54.4 (10.28) | 54.1 (11.07) | 52.6 (11.35) | 51.2 (11.26)

ADVERSE EVENTS:
Time Frame: Up to End-of-Study
Description: End-of-study means 8 weeks after last dose administration. i.e. If patient completed the study, End-of-study visit would be Week 62. If patient could not completed the study, End-of-study visit would be 8 weeks after last dose administration.
Arm/Group | CT-P13 - CT-P13 | CT-P13 - Remicade | Remicade - Remicade | Remicade - CT-P13
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/55 | 0/54 | 0/55
Serious Adverse Events (participants affected / at risk) | 4/56 | 4/55 | 4/54 | 7/55
Other Adverse Events (participants affected / at risk) | 37/56 | 36/55 | 36/54 | 40/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CT-P13 - CT-P13 (N=56) | CT-P13 - Remicade (N=55) | Remicade - Remicade (N=54) | Remicade - CT-P13 (N=55)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abscess intestinal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritoneal tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tuberculous pleurisy (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CT-P13 - CT-P13 (N=56) | CT-P13 - Remicade (N=55) | Remicade - Remicade (N=54) | Remicade - CT-P13 (N=55)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 8 (9) | 5 (7) | 4 (6)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 3 (3) | 3 (3) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 1 (2) | 3 (4) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (4) | 3 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Influenza (Infections and infestations) | 2 (3) | 1 (1) | 1 (1) | 5 (6)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1) | 4 (5) | 3 (3)
Gamma-glutamyltransferase increased (Investigations) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 5 (5) | 5 (5) | 4 (4)
Infusion-related reaction (Injury, poisoning and procedural complications) | 8 (13) | 2 (2) | 5 (7) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1) | 4 (5) | 4 (4)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 4 (4)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 2 (2) | 3 (3)
Pyrexia (General disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No